CLINICAL TRIAL: NCT01404403
Title: Safety Study of the Rapid System for Acute Ischemic Stroke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rapid Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 002-07-01-RR
Record Dates: First submitted 2011-07-26; First posted 2011-07-28 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

ARMS (1):
- Stroke patients (Other)
  Interventions: Device: Rapid System

INTERVENTIONS:
Device: Rapid System

SUMMARY:
This is a safety study of the Rapid System for acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 to <85 years old
* Pre stroke modified Rankin Scale (mRS) of ≤2
* A signed informed consent by patient or a legally acceptable representative

Exclusion Criteria:

* Pre-stroke life expectancy of less than 6 months
* Current participation in another investigational drug or device study
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with Adverse Device Effects (ADEs) Percentage of participants with Adverse Device Effects (ADEs)Percentage | 12 patients

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Hospital, Stockholm, Solna, Sweden